CLINICAL TRIAL: NCT00568451
Title: Releasing the Cancer Patient's Immune System From Down-regulation With Timed Delivery of Standard Chemotherapy
Brief Title: Paclitaxel and Carboplatin or Temozolomide in Treating Patients With Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC057F; P30CA015083 (NIH); MC057F (Other: Mayo Clinic Cancer Center); 06-002547 (Other: Mayo Clinic IRB); NCI-2010-01794 (Registry Identifier: CTRP)
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2014-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Carboplatin; Paclitaxel; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PC (previously treated) (Experimental): Previously chemotherapy treated cohorts: Paclitaxel and Carboplatin (PC)
  Interventions: Drug: carboplatin; Drug: paclitaxel
- PC (chemo naive) (Experimental): Chemotherapy-naive cohorts: Paclitaxel and Carboplatin (PC)
  Interventions: Drug: carboplatin; Drug: paclitaxel
- TMZ (previously treated) (Experimental): Previously chemotherapy treated cohorts: Temozolomide (TMZ)
  Interventions: Drug: temozolomide
- TMZ (chemo naive) (Experimental): Chemotherapy-naive cohorts: Temozolomide (TMZ)
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: carboplatin — AUC=2 intravenously on days 1, 8 and 15. Re-treat every 4 weeks until progression, unacceptable toxicity, or refusal
  Arms: PC (chemo naive); PC (previously treated)
Drug: paclitaxel — 100mg/m^2 intravenously on days 1, 8 and 15. Re-treat every 4 weeks until progression, unacceptable toxicity, or refusal
  Other Names: Taxol
  Arms: PC (chemo naive); PC (previously treated)
Drug: temozolomide — 150mg/m^2 at cycle 1, 200mg/m^2 at cycle 2 and beyond, orally on days 1-5. Re-treat every 4 weeks until progression, unacceptable toxicity, or refusal. One treatment cycle=four weeks
  Other Names: Temodar
  Arms: TMZ (chemo naive); TMZ (previously treated)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving paclitaxel together with carboplatin is more effective than giving temozolomide alone in treating patients with melanoma.

PURPOSE: This phase II trial is studying the side effects and how well giving paclitaxel together with carboplatin or giving temozolomide alone works in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the anti-tumor activity and toxicity profile of timed delivery of conventional paclitaxel and carboplatin (PC) in patients with stage IV melanoma who have received prior chemotherapy for their metastatic disease.
* To assess the anti-tumor activity and toxicity profile of timed delivery of conventional temozolomide (TMZ) chemotherapy in patients with stage IV melanoma who have received prior chemotherapy for their metastatic disease.
* To assess the anti-tumor activity and toxicity profile of timed delivery of conventional PC in patients with stage IV melanoma who have not received prior chemotherapy for their metastatic disease.
* To assess the anti-tumor activity and toxicity profile of timed delivery of conventional TMZ chemotherapy in patients with stage IV melanoma who have not received prior chemotherapy for their metastatic disease.
* To evaluate the changes of T-regulator cells, melanoma-specific functional parameters as a function of time in all four patient cohorts.

OUTLINE: Patients are stratified according to prior chemotherapy for metastatic disease (yes vs no) and scheduled chemotherapy regimen (paclitaxel and carboplatin vs temozolomide).

Beginning at the predicted day of C-reactive peptide (CRP) peak levels, patients receive paclitaxel IV and carboplatin IV on days 1, 8, and 15 OR oral temozolomide alone on days 1-5. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for pharmacological studies. Samples are analyzed for CRP quantification via ELISA; presence and number of circulating blood T-regulator cells via immunophenotyping for CD4/CD25+ and CD4/fox-p3+ T cells; level of functional immunity against melanoma specific antigens (MART-1, tyrosinase, and gp100) and survivin in patients that are HLA-A2+ via intracellular staining; total number of cytotoxic T lymphocytes (CTLs) capable of reacting against melanoma targets via tetramer staining (Becton-Coulter); and quantification of interferon γ-producing, peptide-specific CTLs via multicolor conventional flow cytometry.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic melanoma

  * Stage IV disease
  * Progressive disease
  * No known standard therapy that is potentially curative or proven capable of extending life expectancy exists
* Planning to undergo chemotherapy with paclitaxel and carboplatin OR temozolomide alone for progressive disease
* Measurable disease as defined by RECIST criteria

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mL
* Platelet count ≥ 100,000/mL
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 2.5 x upper limit of normal (ULN)
* AST ≤ 3 x ULN
* Alkaline phosphatase ≤ 3.0 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study therapy
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Active infection
  * NYHA class III or IV congestive heart failure
* No history of other malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix
* Willing to provide research blood samples

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior chemotherapy (patients who received chemotherapy in the metastatic setting)

  * No prior chemotherapy treatment with agents similar to study drugs
* No prior chemotherapy in the metastatic setting (for chemo-naive patients)
* No concurrent enrollment in a different clinical study in which investigational procedures or agents are being used
* No other concurrent investigational agents
* No other concurrent chemotherapy or radiotherapy, including palliative radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve (12) participants with un-resectable stage IV malignant melanoma were enrolled in the study between June 2006 and November 2008 at Mayo Clinic Rochester.
Pre-assignment Details: One patient canceled participation in the trial prior to starting Temozolomide therapy. This patient was excluded from all analysis.
Period: Overall Study
Arm/Group | PC (Previously Treated) | PC (Chemo Naive) | TMZ (Previously Treated) | TMZ (Chemo Naive)
Started | 0 | 0 | 2 | 9
Completed | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 2 | 7
Not completed — Disease Progression | 0 | 0 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PC (Previously Treated) | PC (Chemo Naive) | TMZ (Previously Treated) | TMZ (Chemo Naive) | Total
Number analyzed (Participants) | 0 | 0 | 2 | 9 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 61.5 (14.85) | 63.3 (14.05) | 62.4 (12.97)
Gender [Number; unit: participants]
  Female |  |  | 0 | 3 | 3
  Male |  |  | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States |  |  | 2 | 9 | 11
M Stage [Number; unit: participants] — M stage is based on whether the melanoma has metastasized (spread) to distant organs, which organs it has reached, and on blood levels of a substance called LDH.
  participants
    M1a (skin/subcutaneous tissue/lymph node only) |  |  | 0 | 1 | 1
    M1b (lung) |  |  | 1 | 3 | 4
    M1c (other visceral sites) |  |  | 1 | 5 | 6
Number of Metastatic Sites [Median (Full Range); unit: Sites] |  |  | 2 [2 to 2] | 2 [1 to 5] | 2 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Tumor Status of Either a Complete Response(CR) or Partial Response (PR), According to RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Description: Response that was noted on 2 consecutive evaluations for at least 4 weeks apart.
  CR: Disappearance of all target lesions; PR: At least a 30 percent of decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Target lesions: All measurable lesions up to a maximum of 10 lesions representative of all involved organs.
Time Frame: Every other cycle of therapy (cycle=4 weeks) for the first 6 cycles of treatment
Population: All subjects enrolled, met the eligibility criteria who have signed a consent form and have begun their study treatment were evaluable for response.
Measure: Number; unit: participants
Arm/Group | PC (Previously Treated) | PC (Chemo Naive) | TMZ (Previously Treated) | TMZ (Chemo Naive)
Number analyzed (Participants) | 0 | 0 | 2 | 9
participants |  |  | 0 | 2

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from registration to documentation of disease progression. Disease progression was measured according to the RECIST criteria. Progression: At least a 20 percent increase in the sum of of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Overall: TMZ (Previously Treated) and TMZ (Chemo Naive)
Arm/Group | Overall
Number analyzed (Participants) | 11
Days | 74 [68 to 132]

3. Secondary Outcome: Survival Time
Description: Survival time was defined as the time from registration to death due to any cause.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall
Number analyzed (Participants) | 11
Months | 12.5 [4.5 to NA] — There is not enough events reported to compute 95% CI upper limit.
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; Kaplan-Meier; Median = 12.5, 95% CI 1-sided [lower limit 4.5]

4. Secondary Outcome: Duration of Response for All Evaluable Patients Who Have Achieved an Objective Response
Description: Duration of response was defined as the date at which the participant's objective status was first noted to be either a Complete Response or Partial Response to the date the progression was documented.
Time Frame: up to 2 years
Population: Two complete tumor responses were documented. Both participants have since discontinued the study drug after 35 and 24 cycles respectively, and remain disease-free at 39 and 31.5 months since study entry. There is not enough participants to perform this analysis.
Arm/Group | Overall
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Experienced Changes in Immunologic Profile (CD4/CD25+ Cells, CD4/Fox-p3+ T Cells) Within a Treatment
Description: Time series plot of the number of circulating cells will be constructed. The resulting plots will be visually inspected for trends within and between treatments. For each cell type, a point and an interval estimate of the number of participants (receiving a given treatment) who had at least a 2-fold increase in the number of circulating cells of that type will be constructed using the properties of the binomial distribution.
Time Frame: up to 2 years
Population: There is not enough participants to perform this analysis.
Arm/Group | Overall
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Who Experienced Changes in Immunologic Profile (MART-1, Tyrosinase, and gp100) Within a Treatment
Description: For those patients who are HLA-A2+, the maximum post-treatment levels of MART-1, tyrosinase, and gp100 will be determined. For each of these specific melanoma specific antigens, the number of participants (within a given treatment) who gained or maintained immunity based on the maximum post-treatment level of that specific melanoma specific antigen will be determined.
Time Frame: up to 2 years
Population: There is not enough participants to perform this analysis.
Arm/Group | Overall
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Experienced Changes in Immunologic Profile (IFNγ Producing Peptide Specific CTLs) Within a Treatment
Description: For each patient, a time series plot of the number of IFNγ producing peptide specific CTLs will be constructed. The resulting plots will be visually inspected for trends within and between treatments. A point and an interval estimate of the number of participants (receiving a given treatment) who had at least a 2-fold increase in the number of the number of IFNγ producing peptide specific CTLs will be constructed using the properties of the binomial distribution.
Time Frame: up to 2 years
Population: There is not enough participants to perform this analysis.
Arm/Group | Overall
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | TMZ (Previously Treated) | TMZ (Chemo Naive) | PC (Previously Treated) | PC (Chemo Naive)
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/9 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 8/9 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMZ (Previously Treated) (N=2) | TMZ (Chemo Naive) (N=9) | PC (Previously Treated) (N=0) | PC (Chemo Naive) (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMZ (Previously Treated) (N=2) | TMZ (Chemo Naive) (N=9) | PC (Previously Treated) (N=0) | PC (Chemo Naive) (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 6 (29) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 1 (13) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 0 (0) | 2 (10) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 4 (8) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was stopped prior to achieving its accrual goals due to slow enrollment rate. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes